CLINICAL TRIAL: NCT05224687
Title: Utility Assessment of a Pharmacy-to-Dose Daptomycin Protocol: A Retrospective Cohort Study
Brief Title: Utility Assessment of a Pharmacy-to-Dose Daptomycin
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 068.PHA.2021.A
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Antibiotics Causing Adverse Effects in Therapeutic Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Daptomycin are dosed solely by pharmacists: Daptomycin at two institutions are dosed solely by pharmacists
  Interventions: Other: Retroactive review of patient data of those receiving a dose of daptomycin
- daptomycin protocol is not used and dose by the provider: daptomycin PTD is optional or not utilized at the other institutions.
  Interventions: Other: Retroactive review of patient data of those receiving a dose of daptomycin

INTERVENTIONS:
Other: Retroactive review of patient data of those receiving a dose of daptomycin — A retrospective analysis will be conducted using patient data of those receiving a dose of daptomycin at MCMC, Methodist Dallas Medical Center, Methodist Richardson Medical Center, or Methodist Mansfield Medical Center.

SUMMARY:
A pharmacy-to-dose (PTD) service, also referred to as pharmacy-based dosing, describes an established practice where providers can consult pharmacists for the dosing of various medications. Consulted pharmacists develop a treatment regimen utilizing protocols that are evaluated and approved by the relevant multidisciplinary committees of an institution.

Delegating tasks of therapy monitoring and dose selection to pharmacists resolves providers from this burden and ensures necessary changes are not unnoticed. Daptomycin was a medication that our facility included in PTD because of the required adjustments for renal dysfunction, indication dependent dosing, and its impact on clinical outcomes.

In 2019, our institution approved a PTD daptomycin protocol which allowed pharmacists to select a dose based on provider-selected indications, patient renal function, and body mass index. Pharmacists were also authorized to order creatine phosphokinase (CPK) levels at baseline and every 7 days, if the patient remained on daptomycin. Rounding the dose to the nearest 50 mg or vial size, as deemed appropriate, was also allowed. Daptomycin was one antimicrobial to be added to our growing list of PTD-approved medications. As such, pharmacists were already well acclimated to PTD processes by the time daptomycin was approved for this service.

DETAILED DESCRIPTION:
A pharmacy-to-dose (PTD) service, also referred to as pharmacy-based dosing, describes an established practice where providers can consult pharmacists for the dosing of various medications. Consulted pharmacists develop a treatment regimen utilizing protocols that are evaluated and approved by the relevant multidisciplinary committees of an institution. The Institute for Healthcare Improvement (IHI) recommends implementing pharmacy-based dosing to improve core processes for ordering medications.

Consults for PTD services that require a provider to enter the desired medication and indication have been evaluated in prior studies. This type of consultation requires a clinical or staff pharmacist to implement a patient-specific dosing regimen in addition to ordering of pertinent labs for therapeutic monitoring. Literature on PTD is most prominent regarding pharmacist led services for the dosing and monitoring of vancomycin and aminoglycosides. This is expected because appropriate use of both vancomycin and aminoglycosides relies on ordering and assessment of pharmacokinetic (PK) measurements. As new recommendations for vancomycin dosing and monitoring evolve in complexity, these services are becoming even more valuable. Hospitals with pharmacist-managed vancomycin and aminoglycoside therapy have shown lower drug costs, hearing and renal impairment, and death rates in Medicare patients compared to hospitals without these services.

Other medications that either require renal adjustments, have a narrow therapeutic index, include a wide range of dosing for various indications, or require careful consideration of patient-specific factors are excellent candidates for expanded PTD services. Pharmacists serve as institutions' medication experts and are equipped with knowledge and references needed to apply patient specific characteristics to the selection of a dosing regimen. Medications that require monitoring for the prevention of adverse effects or changes in dosing, often due to the dynamic nature of hospitalized patients' renal function, sometimes go unaddressed. Delegating tasks of therapy monitoring and dose selection to pharmacists resolves providers from this burden and ensures necessary changes are not unnoticed. Daptomycin was a medication that our facility included in PTD because of the required adjustments for renal dysfunction, indication dependent dosing, and its impact on clinical outcomes.

Daptomycin is a cyclic lipopeptide antibiotic that exhibits rapid bactericidal activity against Gram-positive organisms, including various drug resistant isolates of Enterococcus and Staphylococcus. The mechanism does not involve entrance into the bacterial cytoplasm but rather the dissipation of the membrane potential, which occurs through permeable oligomeric lesions in a calcium-dependent fashion. Peak concentration (Cmax)/minimum inhibitory concentration (MIC) and area under the curve (AUC24h)/MIC ratios have been shown in vivo to correlate best with efficacy. Doses of 4 and 6 mg/kg/dose are Food and Drug Administration (FDA)-approved to treat complicated skin and skin structure infections and S. aureus bloodstream infections including right-sided infective endocarditis, respectively. The MICs of daptomycin for Gram-positive cocci differ. Enterococcus faecalis is marked susceptible with MICs ≤ 2 µg/mL; however, strains of Enterococcus faecium display intrinsically higher MICs, and dose-dependent susceptibility based on treatment doses of 8-12 mg/kg/day.

In 2019, our institution approved a PTD daptomycin protocol which allowed pharmacists to select a dose based on provider-selected indications, patient renal function, and body mass index. Pharmacists were also authorized to order creatine phosphokinase (CPK) levels at baseline and every 7 days, if the patient remained on daptomycin. Rounding the dose to the nearest 50 mg or vial size, as deemed appropriate, was also allowed. Daptomycin was one antimicrobial to be added to our growing list of PTD-approved medications. As such, pharmacists were already well acclimated to PTD processes by the time daptomycin was approved for this service.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Have weight and renal function documented prior to daptomycin order entry
* Received at least one dose of daptomycin at any MHS facility

Exclusion Criteria:

* Patients will be excluded if daptomycin was started at an outside facility and their dose was continued during their inpatient stay.

Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving a dose of daptomycin at MCMC, Methodist Dallas Medical Center, Methodist Richardson Medical Center, or Methodist Mansfield Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients receiving appropriate dosing of daptomycin based on indication, weight | July 2019 to October 2021
  Weight in pounds
The primary endpoint is the proportion of patients receiving appropriate dosing of daptomycin based on indication renal function | July 2019 to October 2021
  creatinine clearance

CONTACTS AND LOCATIONS:
Overall Officials: Ronda Akins, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No